CLINICAL TRIAL: NCT00597389
Title: The Efficacy of Early Propranolol Administration at Preventing/Reducing PTSD Symptoms in Child Trauma Victims: Pilot.
Brief Title: Propranolol Administration and Prevention of Child PTSD in Child Trauma Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: Akron Children's Hospital (Other); Ohio Board of Regents (Unknown)
Responsible Party: Douglas L. Delahanty/ Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 04-326
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Posttraumatic Stress Disorders
Keywords: posttraumatic stress disorder; propranolol; inderol; child; trauma; Posttraumatic stress disorders (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): oral solution of propranolol (propranolol HCL 20 mg/5 ml solution) or a liquid placebo twice daily for 10 days (and taper for 5 days; based on Pitman et al, 2002). Dose was calculated as determined by Famularo et al. (1988) to be 2.5 mg/kg/d with a maximum dose of 40 mg bid (Green, 2001).
  Interventions: Drug: Inderol (propranolol)
- 2 (Placebo Comparator): A 25/5ml solution of placebo (a sugar solution that looks and tastes like the propranolol solution)
  Interventions: Drug: Inderol (propranolol)

INTERVENTIONS:
Drug: Inderol (propranolol) — Children ingested a propranolol HCL 20 mg/5 ml solution twice daily for 10 days (and taper for 5 days). Medication was initiated within 12 hours post-trauma. Dose was calculated to be 2.5 mg/kg/d with a maximum dose of 40 mg.
  Other Names: propranolol

SUMMARY:
Twenty-nine pediatric injury patients (ages 10-18) at risk for PTSD were randomly assigned to receive either propranolol or placebo in a double-blind placebo controlled design. Medication was initiated within 12 hours of hospital admission. At 6-weeks, child PTSD symptoms and heart rate (HR) during trauma recall were assessed. We hypothesized that participants who received propranolol would report fewer PTSD symptoms and have lower heart rates than those who received placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants consisted of 15 male and 14 female accidental injury patients aged 10-18 recruited from the emergency department of Akron Children's Hospital. - Eligibility criteria included a Glasgow Coma Scale (GCS) score of 14 or greater (to permit informed consent) and an "at-risk" child score on the STEPP (Winston, Kassam-Adams, Garcia-Espana, Ittenbach, & Cnaan, 2003), a screen for risk of PTSD.

Exclusion Criteria:

* Medication-specific exclusion criteria included hypersensitivity to beta-blockers
* Bradycardia
* Cardiogenic or hypovolemic shock
* Diabetes
* Preexisting heart condition; OR
* Treatment for asthma within the year prior to study entry (per Lacy, Armstrong, Goldman, & Lance, 2002).
* Children were also excluded if they received epinephrine during emergency care or if they sustained any injuries precluding initiation of the propranolol regimen within 12 hours post-trauma.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2004-02; Primary Completion 2005-11 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms with the Clinician Administered PTSD Scale for Children and Adolescents (CAPS-CA) | 6-week follow-up

SECONDARY OUTCOMES:
cardiovascular reactivity during trauma description | at 6-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Delahanty, PhD, Principal Investigator — Kent State University

REFERENCES:
- [Result] The efficacy of early propranolol administration at preventing/reducing PTSD symptoms in child trauma victims: Pilot. Nugent, Nicole Renee; Dissertation Abstracts International: Section B: The Sciences and Engineering, Vol 68(4-B), 2007. pp. 2665.